CLINICAL TRIAL: NCT04652843
Title: Single-center Pathophysiological Study of the Role of Inflammation, Changes in the Intestinal Epithelial Barrier and the Intestinal Microbiota in Parkinson's Disease
Acronym: IBIM-Park
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Despite an extension of the planned duration of inclusion and an enrolled patient number inferior than planned, coordinating investigator considered that it was more reasonable to stop inclusions in order to analyze the data already available
Sponsor: Nantes University Hospital (Other)
Collaborators: France Parkinson Association (Other); Luxia Scientific (Industry); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RC19_0401
Record Dates: First submitted 2020-11-25; First posted 2020-12-03 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Idiopathic REM sleep behavior disorders (Other): Group of 20 Patients with an Idiopathic REM sleep behavior disorder confirmed by video-polysomnography (International Classification of Sleep Disorders-3 criteria), not explained by a pathology (narcolepsy, brainstem injury, neurodegenerative disease)
  Interventions: Procedure: Rectosignoidoscopy; Procedure: Coloscopy
- Beginning Parkinson's disease (Other): Group of 20 patients with Parkinson's Disease which has been progressing for less than 5 years and who have not received dopatherapy
  Interventions: Procedure: Rectosignoidoscopy; Procedure: Coloscopy
- Parkinson's disease state Phase (Other): Group of 20 patients with Parkinson's Disease for more than 5 years
  Interventions: Procedure: Rectosignoidoscopy; Procedure: Coloscopy
- Control (Other): Group of 20 patients undergoing coloscopy for family screening for digestive polyps
  Interventions: Procedure: Coloscopy

INTERVENTIONS:
Procedure: Rectosignoidoscopy — Rectosignoidoscopy for colonic biospsies collection
  Arms: Beginning Parkinson's disease; Idiopathic REM sleep behavior disorders; Parkinson's disease state Phase
Procedure: Coloscopy — Coloscopy for colonic biospsies collection

SUMMARY:
Converging evidence from the literature suggests that digestive inflammation may play a role in the development of Parkinson's disease (PD). The investigators showed in the laboratory in a pilot study that PD patients have digestive inflammation and that the level of inflammation was inversely related to the length of the disease course. This digestive inflammation could be at the origin of an increased intestinal permeability in a subpopulation of parkinsonian patients, cause or consequence of modifications of the intestinal microbiota, thus offering a potential portal of entry for a pathogen according to Braak's theory. To opponents of this theory, it could also reflect the spread of inflammation from the Central nervous System to the Enteral Nervous System (ENS), via the brain-gut axis.

Investigators' hypothesis is that digestive inflammation occurs very early in Parkinson's disease and that it is associated with hyperpermeability of the intestinal epithelial barrier and a change in the intestinal microbiota composition. The investigators propose to study the inflammation markers in the ENS of patients with a pre-motor form of PD (idiopathic Rapid Eye Movement (REM) sleep behavior disorder, n = 20), early-stage PD (<5 years, without dopatherapy, n = 20), more advanced PD (> 5 years, n = 20) and control subjects (n = 20), on colonic biopsies taken during a rectosigmoidoscopy or a coloscopy. Intestinal permeability will be measured by ex-vivo techniques (in a Ussing chamber), the composition of the microbiota will be established by sequencing 16s RNA and the lesional load of phosphorylated alpha-synuclein will be evaluated by immunohistochemistry. All of these parameters will be correlated with clinical data on the severity of PD: duration of development, age, total Unified Parkinson's Disease Rating Scale (UPDRS) motor score and axial sub-score, cognitive tests (Montreal Cognitive Assessment, MoCA), existence of a probable idiopathic REM sleep behavior disorder (REM Sleep Behavior Disorder Screening Questionnaire RBDSQ), olfactory tests, complaint of dysautonomia (SCales for Outcomes in Parkinson's disease - autonomic dysfunction, SCOPA-Aut).

The analysis of inflammation markers, the intestinal barrier and the microbiota could be a first step making it possible to formulate physiopathological hypotheses on the development of PD, to propose predictive biomarkers of the disease and its severity and to design early interventions in the hope of modifying the evolutionary course of the pathological process.

ELIGIBILITY:
Inclusion Criteria:

Parkinson's Disease patients :

* patients with Parkinson's disease according to the criteria of the United Kingdom Parkinson's disease survey brain bank (UKPDSBB)
* aged over 18 years
* who have given their consent to participate in this study

Idiopathic REM sleep behavior disorders patients:

* patients with an Idiopathic REM sleep behavior disorder confirmed by video-polysomnography (International Classification of Sleep Disorders-3 criteria), not explained by a pathology (narcolepsy, brainstem injury, neurodegenerative disease)
* aged over 18 years
* having given their consent to participate in this study

Control:

* patients undergoing coloscopy for family screening for digestive polyps
* aged over 18
* who have given their consent to participate in this study

Exclusion Criteria:

* dementia (MINI MENTAL STATE EXAMINATION score <24)
* history of authenticated colonic disease (inflammatory disease, adenocarcinoma) or functional colopathy in control subjects or having preceded the first signs of Parkinson's Disease or Idiopathic REM sleep behavior disorder for more than 5 years, respectively in Parkinson's Disease and Idiopathic REM sleep behavior disorder patients
* history of prescription of antibiotic treatment, acute gastrointestinal illness or hospitalization for an acute medical pathology or for a surgical procedure in the last month
* anticoagulant treatment or coagulopathy
* pregnant or breastfeeding women, woman not benefiting from effective contraception if of childbearing age
* adults under tutorship, curatorship or under legal protection

For patients with Idiopathic REM sleep behavior disorder:

- presence of Parkinson's Disease according to United Kindom Parkinson's Disease Brain Bank criteria

For control:

* presence of a Parkinson's Disease according to United Kindom Parkinson's Disease Brain Bank criteria
* complaint of nighttime unrest in favor of a probable Idiopathic REM sleep behavior disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
TNF-α | In the three months following the inclusion
  TNF-α in colonic biopsies measured by ELISA

SECONDARY OUTCOMES:
IFN-γ | In the three months following the inclusion
  IFN-γ in colonic biopsies measured by ELISA
IL-6 | In the three months following the inclusion
  IL-6 in colonic biopsies measured by ELISA
IL-1β | In the three months following the inclusion
  IL-1β in colonic biopsies measured by ELISA
IFN-α2 | In the three months following the inclusion
  IFN-α2 in colonic biopsies measured by ELISA
MCP-1 (CCL2) | In the three months following the inclusion
  MCP-1 (CCL2) in colonic biopsies measured by ELISA
IL-8 (CXCL8) | In the three months following the inclusion
  IL-8 (CXCL8) in colonic biopsies measured by ELISA
IL-10 | In the three months following the inclusion
  IL-10 in colonic biopsies measured by ELISA
IL-12p70 | In the three months following the inclusion
  IL-12p70 in colonic biopsies measured by ELISA
IL-17A | In the three months following the inclusion
  IL-17A in colonic biopsies measured by ELISA
IL-18 | In the three months following the inclusion
  IL-18 in colonic biopsies measured by ELISA
IL-23 | In the three months following the inclusion
  IL-23 in colonic biopsies measured by ELISA
IL-33 | In the three months following the inclusion
  IL-33 in colonic biopsies measured by ELISA
Permeability slopes for sulfonic acid | In the three months following the inclusion
  Permeability slopes for sulfonic acid (low molecular weight) and dextran (high molecular weight) measured in a Ussing chamber
Diversity of the intestinal microbiota | In the three months following the inclusion
  Bacterial diversity in each group by genetic sequencing of 16s RNA
Relative abundance of the intestinal microbiota | In the three months following the inclusion
  Relative abundance of different families or genera or bacterial species in each group by genetic sequencing of 16s RNA
Quantification of phosphorylated alpha-synuclein | In the three months following the inclusion
  Presence or absence of inclusion of phosphorylated alpha-synuclein, if presence: quantification (in thioflavin fluorescence intensity and amplification time in minutes)
Duration of progression | At inclusion
  Disease duration of progression as Parkinson's disease clinical severity parameter
Age | At inclusion
  Age as Parkinson's disease clinical severity parameter
Total Unified Parkinson Disease Rating Scale motor score | At inclusion
  Total Unified Parkinson Disease Rating Scale motor score as Parkinson's disease clinical severity parameter
Unified Parkinson Disease Rating Scale axial sub-score | At inclusion
  Unified Parkinson Disease Rating Scale axial sub-score as Parkinson's disease clinical severity parameter
Montreal Cognitive Assessment score | At inclusion
  Montreal Cognitive Assessment score as Parkinson's disease clinical severity parameter
Presence or absence of a probable Idiopathic REM sleep behavior disorders | At inclusion
  Presence or absence of a probable Idiopathic REM sleep behavior disorders (REM Sleep Behavior Disorder Screening Questionnaire score ≥ 5) as Parkinson's disease clinical severity parameter
Olfactory tests | At inclusion
  Olfactory tests (Sniffin 'sticks test score) as Parkinson's disease clinical severity parameter
Scales for Outcomes in Parkinson's Disease - Autonomic Dysfunction score | At inclusion
  Scales for Outcomes in Parkinson's Disease - Autonomic Dysfunction score as Parkinson's disease clinical severity parameter

CONTACTS AND LOCATIONS:
Overall Officials: Laurène LECLAIR-VISONNEAU, MD, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes Universitary Hospital, Nantes, Loire Atlantique, France

IPD SHARING:
Plan to Share IPD: No